CLINICAL TRIAL: NCT04420546
Title: Using Implementation Intentions to Reduce Self-harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Chris Keyworth, Research Fellow, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-8446-15312
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Self-Harm
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (volitional help sheet) (Active Comparator): Participants read a brief statement designed to encourage them to be more physically active ("We want you to plan to increase your level of physical activity"). Participants are presented with a table with two columns and ten rows. Ten 'high risk' situations (temptations) are presented in the left hand column and 10 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted not to be physically active and identifying ways to overcome those temptations had been shown to help people change their behaviour.
  Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from a drop down menu for each critical situation.
  Interventions: Behavioral: Volitional help sheet
- Intervention (volitional help sheet) (Experimental): Participants read a brief statement designed to encourage them to avoid self-harming ("We want you to plan to avoid self-harming"). Participants are presented with a table with two columns and ten rows. Ten 'high risk' situations (temptations) are presented in the left hand column and 10 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to self-harm and identifying ways to overcome those temptations had been shown to help people change their behaviour.
  Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from a drop down menu for each critical situation.
  Interventions: Behavioral: Volitional help sheet

INTERVENTIONS:
Behavioral: Volitional help sheet — Participants are asked to choose from a list of strategies for increasing physical activity
  Arms: Control (volitional help sheet)
Behavioral: Volitional help sheet — Participants are asked to choose from a list of strategies for avoiding self-harm
  Arms: Intervention (volitional help sheet)

SUMMARY:
The aim of the present research is to explore whether a brief intervention based on psychological theory can help people to avoid self-harming. The intervention is the Volitional Help Sheet (VHS), or "IF-THEN" plans, which will be tested in the context of trying to reduce self-harm.

Each participant will be randomly allocated to one of two conditions. The two conditions are: (1) a control condition, and (2) intervention (form multiple implementation intentions from a drop-down menu). The main outcome measure will be reduction in self-harm, which will be self-reported

DETAILED DESCRIPTION:
Background and study aims The purpose of this study is to explore whether a brief intervention based on psychological theory can help people to avoid self-harming. The intervention is the Volitional Help Sheet (VHS), or "IF-THEN" plans, which will be tested in the context of trying to reduce self-harm. An example of an "IF-THEN" plan is "If I feel the urge to self-harm when I want to get relief from a terrible state of mind, Then I will do something else instead of self-harming". IF-THEN plans work by helping people to link a critical situation ("If I am tempted to self-harm when I want to get some attention"), to an appropriate response ("Then I will do something else instead of self-harming").

Implementation intentions (i.e., making if-then plans) are effective at changing behaviour. The investigators have had previous success in using the VHS to reduce self-harm in people recently admitted to hospital for self-harm. The next stage of the research is to explore whether this intervention is acceptable and effective in the population more generally.

Research shows that if people can spot situations in which they may be tempted to self-harm and identify ways of overcoming those situations, they are much more likely to be successful in avoiding self-harming.

Who can participate? Adults aged over 18 years of age, have a history of self-harm, and have good verbal and written understanding of English What does the study involve? The research will involve two phases which aim to examine the acceptability and effectiveness of a brief psychological intervention to reduce self-harm.

Phase 1 Phase 1 involves a wide scale roll out of the VHS, to test the effectiveness of the VHS in reducing self-harm, and to gather feedback about the acceptability of the intervention. YouGov (a survey panel company) will collect the data on behalf of the research team over a period of 6 months (including a baseline and six-month follow-up), and store the data on a secure server, before sending to the research team. The research team at the University of Manchester will conduct and analyse the data. A sample of 1,000 people will take part in Phase 1 and will be randomly allocated to receive either the Volitional Help Sheet (intervention group; to make links between situations and solutions), or a control group (using the same intervention, but for a different behaviour [increasing physical activity]).

Participants will firstly be asked to complete a short series of demographic questions and questions to assess any psychological aspects involved in self-harm. Participants will also be asked about history of self-harm and will be presented with a VHS. Participants in the intervention group will then be asked to construct "IF-THEN plans" for self-harm; participants in the control group will be asked to construct "IF-THEN plans" for increasing physical activity. After participants have been exposed to the VHS, they will be invited to complete a series of questions about their experiences of the VHS and taking part in the study generally. These questions are to assess the feasibility and acceptability of the VHS. All questions will be optional, and participants can choose to skip any should they desire. Likert scale responses and open-ended text fields have been created based on a published framework.

The investigators have gathered some detailed feedback on the VHS from a Patient and Public Involvement and Engagement (PPI/E) group. This group have been specifically trained to provide feedback on research and materials to be used as part of intervention delivery. All members of this group have a history of self-harm. The feedback has been used to ensure the VHS is understandable and sensitive to people's thoughts and emotions. The modified version of the VHS will be implemented in this study.

Participants will be invited to take part in a 6-month follow-up to test the effectiveness of the intervention on recurrence of self-harming. In both the baseline and follow-up questionnaires, YouGov will collect the data on behalf of the research team. YouGov will ensure that all data collected is stored confidentially in accordance with their privacy policy, which participants can view here https://yougov.co.uk/about/terms-combined/#/privacy. Data will be anonymised and sent to the research team at the University of Manchester, where all information will be kept confidential and will conform to the 'Data Protection Act of 1998' with respect to data collection, storage and destruction. Participants' data will be kept separately in secure databases. The participants involved in phase 1 will be recruited as part of a pre-determined sampling frame (developed by YouGov and The University of Manchester), which is intended to be representative of people in the UK who have previously self-harmed.

Phase 2 In between the baseline and follow-up data collected in Phase 1, the investigators will collect an additional round of data on the acceptability of the intervention.

In phase 2 participants will be recruited though online self-harm fora (for example the national Self-harm Network; https://www.nshn.co.uk) and will be invited to complete an online questionnaire. Study adverts will be placed on dedicated pages on each of the fora. The same questionnaire that was used in Phase 1 will be used in Phase 2. As an additional component to phase 2 of the research, participants will be given the option to take part in a short semi-structured telephone interview to discuss the research in further detail. This is entirely optional and if participants do wish to take part, the interview will be conducted at a time and date convenient for them. The interview questions are based on the acceptability questions asked during the questionnaire. If participants wish to take part they will be asked to provide their email address so a member of the research team can contact them to arrange the interview. Based on the findings of Phases 1 and 2 the intervention will be modified and result in a final version of the VHS.

What are the possible benefits and risks of participating? By taking part participants will be helping to understand more about brief interventions to reduce self-harm. By constructing their own "IF-THEN" plans participants are encouraged to construct their own action plans to deal with potential situations where they may be tempted to self-harm.

There are two ethical issues which may arise:

1. Past research indicates that participating in research around self-harm is often a largely positive experience and negative reactions are rare. Our experience running a previous trial using the same intervention as the one in the present application confirms that adverse events are rare. However, there is a low risk of some participants finding the volitional help sheet, which focuses on participants identifying situations where they may feel the urge to self-harm, difficult as it may induce uncomfortable emotions or result in distress.
2. Participants will have a history of self-harm and it is possible that participants will engage in self-harm during or following the study. This risk therefore requires management.

The specific steps taken to address the above are as follows:

1. Steps have been taken to minimize the possible risks identified in this study: All participants will be informed of the possible risk of distress in the Participant Information Sheet. This form will be available to participants online before deciding to take part in the study. Full contact details of the research team will also be provided should participants wish to discuss any queries before they are asked to consent to take part. It will also be suggested to participants that if they feel that taking part in the study will induce significant emotional distress or could increase feelings related to self-harm then they may not want to take part.

   All participants will be informed they do not need to answer any questions they do not wish to, and will be free to withdraw from the study at any time without detriment to themselves. Participants will be advised to withdraw from the study at any point should they become distressed (possibly stopping altogether, or taking a break depending on how the participant wants to proceed).

   Where participants experience significant distress they will be encouraged to speak with their General Practitioner about this at the earliest opportunity.
2. It is reasonable to expect that some participants will engage in self-harm during the course of the study. Due to the participants being able to take part in this study anonymously, the investigators are not able to inform their clinicians. In line with point (1), if participants experience significant distress or emotional discomfort they will be encouraged to speak with their General Practitioner about this to ensure they receive appropriate support and advice. A list of contact numbers of charities and organisations will also be provided as part of the Participant Information Sheet.

In the case that participants indicate to the researcher (for example if a participant phones or emails the researcher) at any point that they plan to seriously harm themselves, a risk and safety plan protocol will be followed (see attached document). This includes a series of steps to determine the level of risk (low-immediate) and appropriate action plans. Action plans include following a safety plan with the participant, providing emergency contact numbers and contacting clinical colleagues and/or emergency services if immediate risk is expressed (in cases where participants have supplied their contact details). These steps may include the need to break confidentiality, by, for example, informing the emergency services. In such cases this breaking of confidentiality would be discussed with participants, unless there is judged a likelihood that this discussion itself could increase risk.

Participants will be informed of the possibility of confidentiality being broken in this manner in the participant information sheet, prior to consent being sought.

All instances of participants signalling either intent/planning of a serious act of self-harm (i.e. a suicide attempt or self-injury liable to require medical intervention) or reporting actual engagement in these behaviours will be treated as a serious adverse event and standard University of Manchester recording practices would be followed (these can be accessed at: https://www.manchester.ac.uk/research/environment/governance/policies-guidelines/).

Where is the study run from?

The University of Manchester (UK)

When is the study starting and how long is it expected to run for?

May 2020 to December 2020

Who is funding the study?

The study is funded by the National Institute for Health Research.

Who is the main contact?

1. Dr Chris Keyworth Chris.keyworth@manchester.ac.uk
2. Prof Christopher J. Armitage Chris.armitage@manchester.ac.uk

Scientific title

Using IF-THEN plans to reduce self-harm

Study hypothesis

Current study hypothesis as of 19/03/2020:

People who form implementation intentions using the volitional help sheet will report reduced self-harm and suicidal ideation at follow-up compared with people in the control condition.

Any effects of the intervention will be mediated principally through increases in automatic motivation and changes in habits.

Study design Mixed methods study. Primary study design Interventional; two-arm randomised controlled trial.

Secondary study design Qualitative study Trial type Prevention Patient information sheet Not available in web format, please use contact details to request a participant information sheet.

Condition Self-harm Intervention

Participants complete a series of questionnaires about their history of self-harm and are then randomly assigned to one of the two conditions:

1. The volitional help sheet includes a list of situations when people might not want to be physically active (e.g., "If I feel the urge to self-harm when I want to get relief from a terrible state of mind") and a list of solutions to overcoming these (e.g., "then I will do something else instead of self-harming"). Participants are asked to make a link (using drop-down menus as part of the online questionnaire) from the situations that are relevant to them to their chosen solutions. They can create as many situation and solution pairs as they want.
2. The control condition includes the same intervention but for a different target behaviour (increasing physical activity).

After 6 months participants are asked the history of self-harm questions to see if the intervention has reduced self-harm.

Intervention type Behavioural Primary outcome measure

1. Non-suicidal self-harm (NSSH) and suicidal ideation and suicide attempts are measured at baseline and 6 months follow-up using three items drawn from the British Psychiatric Morbidity Survey 'Have you ever seriously thought of taking your life, but not actually attempted to do so?' (Suicidal ideation), 'Have you ever made an attempt to take your life, by taking an overdose of tablets or in some other way?' (Suicidal attempt), and 'Have you ever deliberately harmed yourself in any way but not with the intention of killing yourself? (i.e., self-harm)' (NSSH). Response options for all questions are 'Yes' or 'No'. If respondents answer yes to any of the three questions, timing of last episode and frequency will be asked.

Secondary outcome measures

1. Exposure to suicide and mental imagery about death is measured at baseline and follow-up using seven items adapted from those used in the literature previously
2. Capability, opportunity and motivation (based on COM-B model) is measured using the COM questionnaire at baseline and 6 months follow up
3. Habit is measured using the self-reported habit index (automaticity scale) at baseline and 6 months follow up
4. State self-regulation is measured at baseline and 6 months follow up. Items are adapted from those used previously.
5. Frequencies with which critical situations were encountered and appropriate responses were used.

Data analysis plan Randomisation checks The investigators will run tests on all outcome and demographic variables to determine if there are any baseline differences in any of these between conditions: chi square will be used for categorical variables and ANOVA for continuous variables.

The effect of the intervention on frequency of NSSH, suicidal ideation and suicide attempts will be tested using three mixed-measures ANCOVAs with condition (intervention versus control) as the between participants variable and time (baseline versus 6-month follow-up) as the within-participants variable. Planned contrasts will be used to clarify the anticipated time x condition interactions. For each of these three analyses SES, age and gender will be used as covariates.

Three mediation analyses will be conducted using the Hayes mediation model in SPSS with condition (2 levels: intervention versus control) as the independent variable, and (i) NSSH, (ii) suicidal ideation, (iii) suicide attempts as the dependent variables. The investigators will use regression analyses to compute residual scores that will capture any changes between baseline and follow-up. Thus, changes in exposure, impulsivity, habits, self-regulation (awareness of standards, self-monitoring and self-regulatory effort), and COM (capabilities, opportunities and motivations) will be tested as mediators. For each of these three mediation analyses SES, age and gender will be used as covariates.

Moderator analysis will be conducted to identify whether differential effects across the conditions exist depending upon: impulsivity, which is measured using the Barratt impulsiveness scale, anxiety related to COVID-19, which is measured using the Fear of COVID-19 Scale and Impact of Event Scale at baseline. Physical activity will be compared across groups at follow-up using the International Physical Activity Questionnaire (short form).

Scoring the main outcome measures Non-suicidal self-harm (NSSH) and suicidal ideation and suicide attempts NSSH, suicidal ideation and suicide attempts are calculated as binary variables ('yes' or 'no). Frequency of suicidal thoughts will be calculated as continuous variables.

Impulsivity Total score Exposure to suicide and mental imagery about death Exposure to suicide is calculated as a binary variable ('yes' or 'no). Exposure to mental imagery will be calculated as a total score.

COM (capabilities, opportunities and motivations) Each of the items will be analysed separately as these each measure a separate construct.

Self-regulation Mean of the two items for each of three sub-constructs: awareness of standards, self-monitoring, and self-regulatory effort.

Habits Mean of the four items. Frequencies with which critical situations were encountered and appropriate responses were used Total scores Qualitative study For the follow-up qualitative interview component (used specifically in phase 2), thematic analysis will be used to further explore the issues identified in the online questionnaire, and the experiences of using the Volitional Help Sheet (i.e. making "IF-THEN" plans) to reduce self-harm.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Have a history of self-harm
* Good verbal and written understanding of English

Exclusion Criteria:

* Aged under 18 years of age
* No history of self-harm
* Poor verbal and written understanding of English
* Not currently resident of an inpatient facility for mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Non-suicidal self-harm | 6 months
  'Have you ever deliberately harmed yourself in any way but not with the intention of killing yourself? (i.e., self-harm)' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.
Suicidal ideation | 6 months
  'Have you ever seriously thought of taking your life, but not actually attempted to do so?' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.
suicide attempts | 6 months
  'Have you ever made an attempt to take your life, by taking an overdose of tablets or in some other way?' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.

SECONDARY OUTCOMES:
Exposure to suicide and mental imagery about death | 6 months
  Measured at baseline and follow-up using seven items adapted from those used in the literature previously (https://pubmed.ncbi.nlm.nih.gov/26247914/). Calculated as a binary variable ('yes' or 'no). Exposure to mental imagery will be calculated as a total score.
Capability, opportunity and motivation (based on Capability, Opportunity, Motivation-Behaviour model) | 6 months
  Measured using the Capability, Opportunity, Motivation questionnaire (https://pubmed.ncbi.nlm.nih.gov/32314500/). Each of the items (0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.
Habit | 6 months
  Measured using the self-reported habit index (automaticity scale; https://ijbnpa.biomedcentral.com/articles/10.1186/1479-5868-9-102). This consists of four items (each from 1 to 7). Items are scored from 1 to 7, with a higher mean score indicating higher agreement with the statements.
State self-regulation | 6 months
  Items are adapted from those used previously (https://www.tandfonline.com/doi/abs/10.1080/08870440512331317670).
  Mean of the two items for each of three sub-constructs: awareness of standards, self-monitoring, and self-regulatory effort. Items are scored from 1 to 7, with higher scores indicating higher agreement with the statements.
Frequencies with which critical situations were encountered and appropriate responses were used | 6 months
  Frequencies

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

REFERENCES:
- [Background] O'Connor RC, Ferguson E, Scott F, Smyth R, McDaid D, Park AL, Beautrais A, Armitage CJ. A brief psychological intervention to reduce repetition of self-harm in patients admitted to hospital following a suicide attempt: a randomised controlled trial. Lancet Psychiatry. 2017 Jun;4(6):451-460. doi: 10.1016/S2215-0366(17)30129-3. Epub 2017 Apr 20. PMID 28434871
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Biddle L, Cooper J, Owen-Smith A, Klineberg E, Bennewith O, Hawton K, Kapur N, Donovan J, Gunnell D. Qualitative interviewing with vulnerable populations: individuals' experiences of participating in suicide and self-harm based research. J Affect Disord. 2013 Mar 5;145(3):356-62. doi: 10.1016/j.jad.2012.08.024. Epub 2012 Sep 25. PMID 23021191
- [Background] Dhingra K, Boduszek D, O'Connor RC. Differentiating suicide attempters from suicide ideators using the Integrated Motivational-Volitional model of suicidal behaviour. J Affect Disord. 2015 Nov 1;186:211-8. doi: 10.1016/j.jad.2015.07.007. Epub 2015 Jul 29. PMID 26247914
- [Background] O'Connor RC, Rasmussen S, Hawton K. Distinguishing adolescents who think about self-harm from those who engage in self-harm. Br J Psychiatry. 2012 Apr;200(4):330-5. doi: 10.1192/bjp.bp.111.097808. Epub 2012 Mar 8. PMID 22403089
- [Background] Keyworth C, Epton T, Goldthorpe J, Calam R, Armitage CJ. Acceptability, reliability, and validity of a brief measure of capabilities, opportunities, and motivations ("COM-B"). Br J Health Psychol. 2020 Sep;25(3):474-501. doi: 10.1111/bjhp.12417. Epub 2020 Apr 20. PMID 32314500
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Vanaken L, Scheveneels S, Belmans E, Hermans D. Validation of the Impact of Event Scale With Modifications for COVID-19 (IES-COVID19). Front Psychiatry. 2020 Jul 28;11:738. doi: 10.3389/fpsyt.2020.00738. eCollection 2020. PMID 32848918
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: Adult psychiatric morbidity in England, 2007 — http://doc.ukdataservice.ac.uk/doc/6379/mrdoc/pdf/6379_apms_2007_research_report.pdf